CLINICAL TRIAL: NCT03102346
Title: A Perspective Randomized Controlled Clinical Trial to Investigate the Effect of Home-based Cardiac Rehabilitation Monitored by Mobile Phone Interaction on Exercise Capacity and One-year Clinical Outcome in Chinese Revascularized Patients
Brief Title: efficAcy and Safety of Home-baSed Cardiac rehabIlitation in ChineSe Revascularized patienTs
Acronym: ASSIST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yun Dai Chen, Director, Head of Cardiology, Principal Investigator, Clinical Professor, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S2016-142-01
Record Dates: First submitted 2017-03-25; First posted 2017-04-05 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Coronary Artery Disease
Keywords: cardiorespiratory fitness; coronary artery disease; cardiac rehabilitation; remote control; major adverse cardiac and cerebrovascular events
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based Cardiac Rehabilitation group (Experimental): remote instructed exercise training at home
  Interventions: Other: home-based cardiac rehabilitation
- routine group (No Intervention): no instructed exercise training

INTERVENTIONS:
Other: home-based cardiac rehabilitation — The exercise training includes aerobic exercise (fast walking or cycling ,30-40 minutes per day,5-6 times a week), stretching exercise (15 minutes every time, 5-6 times a week), and resistance and balance training (each of 15 minutes every time, twice to 3 times a week).
  Other Names: exercise training at home
  Arms: Home-based Cardiac Rehabilitation group

SUMMARY:
Home-based CR (HBCR) was reported to improve the clinical outcomes of coronary artery disease (CAD) patients. There is no data published to investigate whether HBCR is also effective for Chinese CAD patients who have been revascularized.

This trial was designed to investigate the safety and efficacy of CR program at home for Chinese patients who underwent PCI (Percutaneous Coronary Intervention) procedure. This is a multicenter, randomized, controlled and observational study.

DETAILED DESCRIPTION:
Numerous studies have revealed that cardiac rehabilitation (CR) after myocardial Cardiac rehabilitation (CR) after revascularization results in better clinical outcomes, and have been strongly recommended for patients with coronary artery disease. In China, as compared to the exponential increase of PCI (Percutaneous Coronary Intervention) volume, only a very small amount of hospitals are able to develop CR programs. There is no large-scale study to explore the feasible CR pattern either. Home-based CR might be more favorable and practical for so many Chinese revascularized coronary artery disease (CAD) patients due to its feasibility and flexibility as well as low medical cost.

This trial was designed to investigate the safety and efficacy of CR program at home for Chinese patients who underwent PCI procedure. This is a multicenter, randomized, controlled and observational study. The efficacy and safety of Home-based CR (HBCR) in revascularized patients will be evaluated through observation of its clinical characteristics and safety indicators. The study will involve 14 sites nationwide, with an expected sample size of 2,000 followed up for 12 months. The primary endpoints is the incidence of composite major adverse cardiac and cerebrovascular events (MACCE,death from any cause, nonfatal myocardial infarction, revascularization, stroke).Secondary endpoints are defined as decrease of hospitalization due to refractory angina pectoris，the improvements of cardiorespiratory fitness,life quality,as well as angina pectoris.

The subjects will be randomized into 2 different groups, HBCR group and control group. After comprehensive evaluation, the orders from CR staff will be given. Besides the routine health education in both groups, the subjects in HBCR group will be further introduced the instructions of exercise training. The effect of HBCR on cardiorespiratory fitness, improvement of angina, cardiac function, quality of life, levels of anxiety and depression, as well as risk factor profile will also be evaluated. The investigators also aim to explore the factors which influence the adherence of subjects to our HBCR program.

ELIGIBILITY:
Inclusion Criteria:

all of them

1. age range from 30 to 80.
2. coronary artery disease,revascularized with stent deployment.
3. New York Heart Association (NYHA) classification Class I-III.
4. Good cognitive level.
5. Ability to perform aerobic exercise.
6. Understand be able to use a mobile smart phone by himself or with help of family members.
7. Signature of informed consent. The informed consent will be valid for the duration of the trial or until the subject withdraws.

Exclusion Criteria (Enrollment):

1. Presence of malignant arrhythmias such as ventricular fibrillation outside the acute phase of Acute myocardial infarction (AMI) (> 24 h after AMI), ventricular tachycardia, Atrioventricular block of 2nd degree and 3rd degree, Atrial fibrilation (FA) in patients with Wolf Parkinson White, fibrillation or paroxysmal atrial flutter with response ventricular quickly and hemodynamic deterioration, premature ventricular contractions increases during exertion, paroxysmal supraventricular tachycardia uncontrolled.
2. Hypotensive response to exercise.
3. acute myocardial infarction within 2 weeks
4. Poorly controlled hypertension baseline,hyperglycemia,respiratory failure.
5. severe pulmonary hypertension
6. acute phase of heart failure
7. Pathology of musculoskeletal, neurological or breathing that impair the ability of prolonged ambulation.
8. Pregnant women.
9. Subjects unable to give informed consent.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2017-11-09 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
MACCE(death, nonfatal myocardial infarction, revascularization, stroke) | during 12 months
  defined as the incidence of composite MACCE.

SECONDARY OUTCOMES:
improvement of hospitalization due to refractory angina pectoris | during 12 months
  improvement of hospitalization due to refractory angina pectoris which need to be treated in hospital
improvement of cardiorespiratory fitness | during 12 months
  peak oxygen uptake adjusted by body weight measured by cardiopulmonary exercise test
improvement of life quality | during 12 months
  measured by medical outcomes study 36-item short form health survey
improvement of angina pectoris | during 12 months
  measured by Seattle Angina Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Yundai Chen, MD,PHD, Principal Investigator — Director of department of Cardiology, Chinese PLA General Hospital
Locations (1):
- the First People's Hospital of Yunnan Province, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DeBusk RF, Miller NH, Parker KM, Bandura A, Kraemer HC, Cher DJ, West JA, Fowler MB, Greenwald G. Care management for low-risk patients with heart failure: a randomized, controlled trial. Ann Intern Med. 2004 Oct 19;141(8):606-13. doi: 10.7326/0003-4819-141-8-200410190-00008. PMID 15492340
- [Background] Haskell WL, Alderman EL, Fair JM, Maron DJ, Mackey SF, Superko HR, Williams PT, Johnstone IM, Champagne MA, Krauss RM, et al. Effects of intensive multiple risk factor reduction on coronary atherosclerosis and clinical cardiac events in men and women with coronary artery disease. The Stanford Coronary Risk Intervention Project (SCRIP). Circulation. 1994 Mar;89(3):975-90. doi: 10.1161/01.cir.89.3.975. PMID 8124838
- [Background] Froelicher V, Jensen D, Genter F, Sullivan M, McKirnan MD, Witztum K, Scharf J, Strong ML, Ashburn W. A randomized trial of exercise training in patients with coronary heart disease. JAMA. 1984 Sep 14;252(10):1291-7. PMID 6381770
- [Background] Newton M, Mutrie N, McArthur JD. The effects of exercise in a coronary rehabilitation programme. Scott Med J. 1991 Apr;36(2):38-41. doi: 10.1177/003693309103600203. PMID 1853191
- [Background] Conraads VM, Van Craenenbroeck EM, Pattyn N, Cornelissen VA, Beckers PJ, Coeckelberghs E, De Maeyer C, Denollet J, Frederix G, Goetschalckx K, Hoymans VY, Possemiers N, Schepers D, Shivalkar B, Vanhees L. Rationale and design of a randomized trial on the effectiveness of aerobic interval training in patients with coronary artery disease: the SAINTEX-CAD study. Int J Cardiol. 2013 Oct 9;168(4):3532-6. doi: 10.1016/j.ijcard.2013.05.007. Epub 2013 May 24. PMID 23711446
- [Background] Soga Y, Yokoi H, Amemiya K, Iwabuchi M, Nobuyoshi M. Safety and efficacy of exercise training after coronary stenting in patients with stable coronary artery disease. Circ J. 2011;75(10):2379-86. doi: 10.1253/circj.cj-11-0470. Epub 2011 Jul 28. PMID 21799272
- [Background] Perez-Terzic CM. Exercise in cardiovascular diseases. PM R. 2012 Nov;4(11):867-73. doi: 10.1016/j.pmrj.2012.10.003. PMID 23174552